CLINICAL TRIAL: NCT05736224
Title: Assessing a Natural Product Plus Bioadhesive Nanoparticle (BNP) Sunscreen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2000033876; 2P50CA121974-11A1 (NIH)
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Results first posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms | interventions — Sunscreening Agents; Ultraviolet Rays

STUDY DESIGN:
Intervention Model Description: Within subject design where participant serves as own control.
Who Masked: Outcomes Assessor
Masking Description: Laboratory technicians will be blinded to treatment of samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sunscreen (Experimental): Portion of skin covered by sunscreen. There are 3 different formulations of sunscreen (Formulation 1, Formulation 2, Formulation 3)
  Interventions: Drug: Sunscreen; Other: UV Light
- No treatment control (Other): Portion of skin not covered by sunscreen.
  Interventions: Other: UV Light

INTERVENTIONS:
Drug: Sunscreen — The sunscreen contains bioadhesive nanoparticles (BNP) encapsulating avobenzone and octocrylene plus the non-toxic natural products diosmin, ferulic acid, cytisine and trans-resveratrol.
  Arms: Sunscreen
Other: UV Light — UV light to the correct sites, and the Multiport 610 solar simulator used to deliver 1 MED UVR to the appropriate subsites.

SUMMARY:
The primary objective of this study is to evaluate the effects of a novel sunscreen formulation by assessing the extent of ultraviolet radiation (UVR)-induced direct and indirect cellular and DNA damage to human skin, in the presence vs absence of the sunscreen, in a population of healthy adults with fair skin (Fitzpatrick Scale type I, II or III).

DETAILED DESCRIPTION:
Skin cancer is the most commonly diagnosed malignancy in the USA and ultraviolet radiation (UVR) exposure is the major environmental risk factor for skin cancer development. Currently available sunscreens utilize UVR filters that, while absorbing UVR energy, have been shown to induce ROS, resulting in oxidative DNA damage after UVR exposure. Organic sunscreen actives have also been shown to penetrate into the skin, raising direct toxicity, as well as irritant and photoallergic concerns. Further systemic absorption may result in additional health risks such as endocrine disruption. Novel sunscreens that more safely prevent both direct and indirect DNA damage are needed.

The study team have produced a bioadhesive nanoparticle (BNP) sunscreen designed to keep organic UVR filters from penetrating into the skin and have incorporated non-toxic natural products into this sunscreen to further safely boost UVR absorbing capacity and reduce oxidative, indirect DNA damage. This study will test the capacity of this sunscreen to prevent direct and indirect cellular and DNA damage in human skin exposed to UVR.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Women of child-bearing potential must have negative urine pregnancy test
* In good general health as evidenced by medical history
* Fair skinned with Fitzpatrick Scale skin types I, II or III using the following Skin Type and Sunburn and Tanning History (based on the first 30-45 minutes of sun exposure after a winter season of no sun exposure):
* I always burns easily; never tans (sensitive)
* II always burns easily; tans minimally (sensitive)
* III burns moderately; tans gradually (light brown) (normal)

Exclusion Criteria:

* Individuals with active or a history of dermatological disorders-psoriasis, rosacea, eczema, vitiligo, lupus, dermatomyositis, etc
* Individuals known to be subject to any abnormal responses to sunlight, such as phototoxic or photoallergic response.
* Current use of medication (topical or systemic) that is known to produce abnormal sunlight responses.
* History of skin cancer (such as basal cell carcinoma, squamous cell carcinoma, melanoma)
* Family history of melanoma
* Presence of sunburn, suntan, scars, active dermal lesions or uneven skin tone on the test site.
* Skin type falling under the Fitzpatrick Scale skin types IV, V or VI using the following Skin Type and Sunburn and Tanning History (based on the first 30-45 minutes of sun exposure after a winter season of no sun exposure):
* IV Burns minimally; always tans well (moderate brown) (normal)
* V Rarely burns; tans profusely (dark brown) (insensitive)
* Use of sunscreen within the last week on the test site area (such that UV filter penetration may confound results)
* Febrile illness within 48 hours.
* Women with a positive urine pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Girardi, MD, FAAD, Principal Investigator — Evans Professor of Dermatology; Director, Residency Program, Dermatology
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results published from this study, after deidentification (text, tables, figures, and appendices), will be made available to researchers who provide a methodologically sound proposal. Proposals should be directed to michael.girardi@yale.edu.
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Access will be given to researchers who provide a methodologically sound proposal. Proposals should be directed to michael.girardi@yale.edu. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunscreen and no Suncreen (All Participants): All participants will have biopsies from a portion of skin with sunscreen applied and a portion of skin without sunscreen applied
Period: Overall Study
Arm/Group | Sunscreen and no Suncreen (All Participants)
Started | 30
Formulation 1 | 8
Formulation 2 | 14
Formulation 3 | 8
Completed | 29
Not Completed | 1
Not completed — Excluded from analysis because processed biopsy sample was inadequate for analysis | 1

BASELINE CHARACTERISTICS:
Population: Race/ethnicity was not collected. Subjects were screened by skin type.
Arm/Group | Sunscreen and no Suncreen (All Participants)
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30
Skin Type (Fitzpatrick) [Count of Participants; unit: Participants] — Fitzpatrick Skin Type I: Pale white skin, blue/green eyes, blond/red hair; Always burns, does not tan
  Fitzpatrick Skin Type II: Fair skin, blue eyes; Burns easily, tans poorly
  Fitzpatrick Skin Type II/III: Between II and III
  Fitzpatrick Skin Type III: Darker white skin; Tans after initial burn
  Participants
    Fitzpatrick Type I | 1
    Fitzpatrick Type II | 20
    Fitzpatrick Type II/III | 2
    Fitzpatrick Type III | 7

OUTCOME MEASURES:

1. Primary Outcome: DNA Damage Level by Cyclobutane Pyrimidine Dimer (CPD) Measurement
Description: Ultraviolet radiation (UVR) exposure are indicative of direct DNA damage. DNA will be prepared and assayed by ELISA for quantification of CPDs. CPDs measured in samples obtained immediately after UVR exposure are indicative of direct DNA damage. DNA from skin biopsies was used to quantify the level of DNA damage, represented by CPD levels detected by enzyme-linked immunosorbent assay (ELISA)
Time Frame: 5 minutes after UVR exposure
Population: Test Sites were delineated on the subjects upper inner arm, then either No sunscreen was applied, or the Test Sunscreen was applied 1 time at the FDA prescribed level (2 mg/cm2) and dried for 15 minutes before UVR exposure. The test sites were biopsied 5 minutes and 4 hours after UVR exposure. Two biopsies (one with sunscreen and one without) were taken per participant.
Measure: Mean (Standard Error); unit: Optical Density Units
Units Other Than Participants: biopsies
Groups:
- Sunscreen Formulation 1; Sunscreen Formulation 2; Sunscreen Formulation 3: Two biopsies were taken per participant: one from portion of skin covered by sunscreen and one where no sunscreen was applied.
  Sunscreen: The sunscreen contains bioadhesive nanoparticles (BNP) encapsulating avobenzone and octocrylene plus the non-toxic natural products diosmin, ferulic acid, cytisine and trans-resveratrol.
  UV Light: UV light to the correct sites, and the Multiport 610 solar simulator used to deliver 1 MED UVR to the appropriate subsites.
Arm/Group | Sunscreen Formulation 1 | Sunscreen Formulation 2 | Sunscreen Formulation 3
Number analyzed (Participants) | 8 | 13 | 8
Number analyzed (biopsies) | 16 | 26 | 16
Optical Density Units
  No sunscreen: number analyzed (biopsies) | 8 | 13 | 8
  No sunscreen | 2.48 (0.15) | 2.18 (0.14) | 2.64 (0.09)
  Sunscreen: number analyzed (biopsies) | 8 | 13 | 8
  Sunscreen | 1.14 (0.26) | 0.33 (0.07) | 1.24 (0.19)
Statistical Analysis 1: Comparison: Sunscreen Formulation 1; Test type: Superiority; p = 0.003, t-test, 2 sided — No sunscreen compared to test sunscreen

2. Primary Outcome: DNA Damage Level by Cyclobutane Pyrimidine Dimer (CPD) Measurement
Description: as for outcome 1
Time Frame: 4 hours after UVR exposure
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Optical Density Units
Units Other Than Participants: biopsies
Arm/Group | Sunscreen Formulation 1 | Sunscreen Formulation 2 | Sunscreen Formulation 3
Number analyzed (Participants) | 8 | 13 | 8
Number analyzed (biopsies) | 16 | 26 | 16
Optical Density Units
  No sunscreen: number analyzed (biopsies) | 8 | 13 | 8
  No sunscreen | 2.41 (0.21) | 2.07 (0.14) | 2.42 (0.08)
  Sunscreen: number analyzed (biopsies) | 8 | 13 | 8
  Sunscreen | 1.03 (0.26) | 0.24 (0.05) | 0.92 (0.23)

3. Primary Outcome: Detectable DNA Strand Breaks
Description: Formalin fixed paraffin embedded skin stained with anti-gH2AX to identify keratinocytes with DNA strand breaks. Indirect, oxidative DNA damage may result in DNA strand breaks that can be visualized by microscopic analysis after staining for gH2AX, which builds up within cells with DNA strand break.
Time Frame: 5 minutes after UVR exposure
Population: as for outcome 1
Measure: Mean (Standard Error); unit: fluorescence units
Units Other Than Participants: biopsies
Arm/Group | Sunscreen Formulation 1 | Sunscreen Formulation 2 | Sunscreen Formulation 3
Number analyzed (Participants) | 8 | 13 | 8
Number analyzed (biopsies) | 16 | 26 | 16
fluorescence units
  No sunscreen (normalized): number analyzed (biopsies) | 8 | 26 | 16
  No sunscreen (normalized) | 0 (0) | 0 (0) | 0 (0)
  Sunscreen (normalized): number analyzed (biopsies) | 8 | 26 | 16
  Sunscreen (normalized) | 0 (0) | 0 (0) | 0 (0)

4. Primary Outcome: Number of DNA Strand Breaks
Description: as for outcome 3
Time Frame: 4 hours after UVR exposure
Population: as for outcome 1
Measure: Mean (Standard Error); unit: fluorescence units
Units Other Than Participants: biopsies
Arm/Group | Sunscreen Formulation 1 | Sunscreen Formulation 2 | Sunscreen Formulation 3
Number analyzed (Participants) | 8 | 13 | 8
Number analyzed (biopsies) | 16 | 26 | 16
fluorescence units
  No sunscreen: number analyzed (biopsies) | 8 | 13 | 8
  No sunscreen | 0 (0) | 0 (0) | 0 (0)
  Sunscreen: number analyzed (biopsies) | 8 | 13 | 8
  Sunscreen | 0 (0) | 0 (0) | 0 (0)

5. Primary Outcome: Cellular Damage
Description: Formalin fixed paraffin embedded skin stained with anti-3-nitrotyrosine to identify cellular damage. ROS and high energy triplet state species can result in nitration of tyrosine residues of cellular proteins. This type of damage can be visualized by microscopic visualization of 3-nitrotyrosine.
Time Frame: 5 minutes after UVR exposure
Population: as for outcome 1
Measure: Mean (Standard Error); unit: fluorescence units
Units Other Than Participants: biopsies
Arm/Group | Sunscreen Formulation 1 | Sunscreen Formulation 2 | Sunscreen Formulation 3
Number analyzed (Participants) | 8 | 13 | 8
Number analyzed (biopsies) | 16 | 26 | 16
fluorescence units
  No sunscreen: number analyzed (biopsies) | 8 | 13 | 8
  No sunscreen | 0 (0) | 0 (0) | 0 (0)
  Sunscreen: number analyzed (biopsies) | 8 | 13 | 8
  Sunscreen | 0 (0) | 0 (0) | 0 (0)

6. Primary Outcome: Cellular Damage
Description: as for outcome 5
Time Frame: 4 hours after UVR exposure
Population: as for outcome 1
Measure: Mean (Standard Error); unit: fluorescence units
Units Other Than Participants: biopsies
Arm/Group | Sunscreen Formulation 1 | Sunscreen Formulation 2 | Sunscreen Formulation 3
Number analyzed (Participants) | 8 | 13 | 8
Number analyzed (biopsies) | 16 | 26 | 16
fluorescence units
  No sunscreen: number analyzed (biopsies) | 8 | 13 | 8
  No sunscreen | 0 (0) | 0 (0) | 0 (0)
  Sunscreen: number analyzed (biopsies) | 8 | 13 | 8
  Sunscreen | 0 (0) | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Sunscreen and no Suncreen (All Participants)
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/24/NCT05736224/Prot_SAP_001.pdf
  • Informed Consent Form (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/24/NCT05736224/ICF_000.pdf